CLINICAL TRIAL: NCT04539587
Title: Sexual Quality of Life in Women During the First Year of Adjuvant Hormonal Treatment for Breast Cancer: a Prospective Longitudinal Study
Brief Title: Sexual Quality of Life in Women During the First Year of Adjuvant Hormonal Treatment for Breast Cancer.
Acronym: CUPIDON
Status: Completed | Type: Observational
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Other Study IDs: PROICM 2018-05 BCU
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2020-08

CONDITIONS: Breast Cancer; Cancer; Quality of Life
Keywords: breast cancer; hormonotherapy; women; quality of life
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adjuvant hormonal therapy for breast cancer: Women more than 18 years old, with hormone receptor-positive early BC, with completed surgery as well as chemotherapy and/or radiotherapy, if indicated, and had begun their hormonal therapy for less than 6 months.
  Interventions: Other: Quality of life

INTERVENTIONS:
Other: Quality of life — The patient will receive the following questionnaires to be completed :
  EORTC QLQ-C30 EORTC QLQ-BR23 EORTC SHQ-C22

SUMMARY:
Breast cancer is the most common cancer in women worldwide. Hormonal therapy is one of the major treatments for hormone receptor positive breast tumors. It is prescribed to 70% of breast cancer patients. Hormonal therapy can be responsible for sexual dysfunction induced by hormonal changes. Extended adjuvant hormonal therapy over 5 years increases these adverse effects.

According to the third "Plan Cancer" (2014-2019), sexual dysfunction prevention and screening must be systematic as an integral part of supportive care. Nevertheless, sexual quality of life remains too rarely considered.

In this study, the investigator propose to evaluate sexual quality of life of women less than 51 years old during the adjuvant endocrine therapy for localized breast cancer. The investigator also intend to collect the supportive measures or interventions used by women to overcome sexual dysfunction. Finally, this study aims to evaluate the need for sexual trouble specific management and acceptability of different methods.

This project is a hot topic as the interest for oncosexuality is growing, and the need for specific management is increasing with still insufficient access to specific care.

DETAILED DESCRIPTION:
Breast cancer (BC) is the most common cancer in women worldwide, affecting approximately one in eight women during her lifetime in Western countries. (chiffres Globocan). Approximately two thirds of BC are hormone receptor-positive and the multimodal treatment will therefore include hormone therapy during 5 years or even longer (Burstein et al. 2019).

Many studies have described a wide range of disruptions in day to day living after breast cancer diagnosis and treatment. These physical, psychological and social concerns for the patients, related to the disease and its treatment, are now recognized as important outcomes in clinical trials and are evaluated in standardized Health-related quality of life (HRQL) questionnaires like the general EORTC QLQ-C30 dedicated to all cancer patients (Aaronson et al. 1993) or the EORTC QLQ-BR23 dedicated to breast cancer patients (Sprangers et al. 1996).

Sexual dysfunction is frequent during and after treatment for breast cancer (Ananth et al. 2003; Krychman et al. 2006; Pup et al. 2019) and is not specifically evaluated in these general HRQL questionnaires. Recently, the EORTC SHQ-C22 has been developed as a standardized instrument to evaluate sexual quality of life (QoL) in cancer patients to address and evaluate in more detail the sexual dysfunction related to the disease and the treatment(Oberguggenberger et al. 2018).

A prospective longitudinal assessment is conduted of the sexual functioning of women during the first year of adjuvant hormonal therapy using global HRQL questionnaires as well as the new SHQ-C22 questionnaire specifically dedicated to sexual QoL for cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Female age ≥ 18 years old
* Patient with non-metastatic early breast cancer,
* Patient undergoing adjuvant hormonal therapy
* Patient who has been treated by surgery, with or without chemotherapy and/or radiotherapy.
* Patient being currently sexually active.
* Patient who agreed, after receiving information, to participate to the study.

Exclusion Criteria:

* - Patient who refused to participate to this study or is unable to fulfill a questionnaire,
* Patient not affiliated to the French social security system,
* Subject under tutelage, curatorship or safeguard of justice,
* Patient in an emergency situation,
* Patient whose regular monitoring is impossible for psychological, family, social or geographical reasons,
* Pregnant and / or breastfeeding woman.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients were minimum 18 years old, had hormone receptor-positive early BC, had all completed surgery as well as chemotherapy and/or radiotherapy, if indicated, and had begun their hormonal therapy for less than 6 months.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Sexual quality of life: EORTC SHQ-C22 questionnaire | At the inclusion, at day 1
  Sexual quality of life assessed by the EORTC SHQ-C22 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Véronique D'HONDT, MD, Study Chair — Institut Régional du Cancer de Montpellier (ICM)
Locations (1):
- Institut régional du Cancer de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cavalheiro JA, Bittelbrunn A, Menke CH, Biazus JV, Xavier NL, Cericatto R, Schuh F, Pinheiro CV, Passos EP. Sexual function and chemotherapy in postmenopausal women with breast cancer. BMC Womens Health. 2012 Sep 11;12:28. doi: 10.1186/1472-6874-12-28. PMID 22963155
- [Background] Dow J, Kennedy Sheldon L. Breast Cancer Survivors and Sexuality: A Review of the Literature Concerning Sexual Functioning, Assessment Tools, and Evidence-Based Interventions. Clin J Oncol Nurs. 2015 Aug;19(4):456-61. doi: 10.1188/15.CJON.456-461. PMID 26207711
- [Background] Frechette D, Paquet L, Verma S, Clemons M, Wheatley-Price P, Gertler SZ, Song X, Graham N, Dent S. The impact of endocrine therapy on sexual dysfunction in postmenopausal women with early stage breast cancer: encouraging results from a prospective study. Breast Cancer Res Treat. 2013 Aug;141(1):111-7. doi: 10.1007/s10549-013-2659-y. Epub 2013 Aug 14. PMID 23942873
- [Background] Hummel SB, van Lankveld JJDM, Oldenburg HSA, Hahn DEE, Kieffer JM, Gerritsma MA, Kuenen MA, Bijker N, Borgstein PJ, Heuff G, Lopes Cardozo AMF, Plaisier PW, Rijna H, van der Meij S, van Dulken EJ, Vrouenraets BC, Broomans E, Aaronson NK. Efficacy of Internet-Based Cognitive Behavioral Therapy in Improving Sexual Functioning of Breast Cancer Survivors: Results of a Randomized Controlled Trial. J Clin Oncol. 2017 Apr 20;35(12):1328-1340. doi: 10.1200/JCO.2016.69.6021. Epub 2017 Feb 27. PMID 28240966